CLINICAL TRIAL: NCT01626755
Title: Prevention of Phantom Limb Pain After Transtibial Amputation (PLATA) - Randomized, Double-blind, Controlled, Multi-center Trial Comparing Optimized Intravenous Pain Control vs Optimized Intravenous Pain Control Plus Nerve Block.
Brief Title: Prevention of Phantom Limb Pain After Transtibial Amputation
Acronym: PLATA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and recruitment.
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: European Society of Anaesthesiology (Other)
Responsible Party: Principal Investigator, Philipp Lirk, Attending Anesthesiologist, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLATA
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Phantom Limb Pain; Chronic Pain; Prevention
Keywords: Phantom limb pain; Chronic pain; Amputation; Peripheral vascular disease
MeSH Terms: conditions — Phantom Limb; Chronic Pain; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nerve block (Experimental): Optimized intravenous pain treatment during surgery and for 7 days postoperatively.
  Definition: strong opioid patient-controlled analgesia, non-opioids, ketamine intravenously.
  Sciatic nerve block: infusion of local anesthetic.
  Interventions: Procedure: Sciatic name block
- Control (Active Comparator): Optimized intravenous pain treatment during surgery and for 7 days postoperatively.
  Definition: strong opioid patient-controlled analgesia, non-opioids, ketamine intravenously.
  Sciatic nerve block: saline infusion.
  Interventions: Procedure: Sciatic name block

INTERVENTIONS:
Procedure: Sciatic name block — Ultrasound-guided sciatic nerve block.

SUMMARY:
Phantom limb pain following amputation is a major problem. Current evidence how to best prevent phantom limb pain is equivocal because previous trials have included small numbers of patients, and tested heterogeneous patient collectives. There is some evidence that optimized perioperative pain control is effective in preventing phantom limb pain, but the potential added role of regional anesthesia has not been defined.

Objective:

The Aim of this study is to test the hypothesis that sciatic nerve block decreases the point prevalence of phantom limb pain 12 months after transtibial amputation for peripheral vascular disease compared to optimized intravenous pain therapy.

Study design:

Randomized, prospective, double-blind (patient, physician, statistician) clinical trial. All patients will receive standard optimized intravenous anesthesia and analgesia (opiate patient-controlled analgesia (PCA), intravenous ketamine). Patients in the intervention group will receive additional infusion of local anesthetic via a sciatic nerve catheter placed under ultrasound guidance.

Main outcome of this study:

Point prevalence of chronic phantom limb pain after 12 months.

DETAILED DESCRIPTION:
Rationale:

Phantom limb pain following amputation is a major clinical problem. Current evidence how to best prevent phantom limb pain is equivocal because previous trials have included small numbers of patients, and tested heterogeneous patient collectives. There is some evidence that optimized perioperative pain control is effective in preventing phantom limb pain, but the potential added role of regional anesthesia has not been defined.

Objective:

The Aim of this study is to test the hypothesis that sciatic nerve block decreases the point prevalence of phantom limb pain 12 months after transtibial amputation for peripheral vascular disease compared to optimized intravenous pain therapy.

Study design:

Randomized, prospective, double-blind (patient, physician, statistician) clinical trial. All patients will receive standard optimized intravenous anesthesia and analgesia (opiate patient-controlled analgesia (PCA), intravenous ketamine). Patients in the intervention group will receive additional infusion of local anesthetic via a sciatic nerve catheter placed under ultrasound guidance.

Study population:

Patients undergoing elective transtibial amputation for peripheral vascular disease at one of the participating centres, ASA status II to IV.

Intervention:

Infusion of local anesthetic via sciatic nerve catheter placed under ultrasound guidance.

Main study parameter/endpoint:

Point prevalence of chronic phantom limb pain after 12 months.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

All patients, regardless of group allocation, will receive optimalized intravenous pain treatment. The aim of this study is to assess whether additional regional anesthesia (ultrasound-guided sciatic nerve block) can decrease the incidence of phantom limb pain. The working hypothesis is that patients undergoing intervention treatment (optimized intravenous therapy plus nerve block) are expected to feature a decreased incidence of phantom limb pain at 12 months, in addition to improved perioperative analgesia.

The administration of both optimalized intravenous pain treatment and peripheral nerve blockade is routine clinical practice for many procedures on the lower leg, including amputation. The risk of this intervention can be described as very low. In control patients, the sciatic catheter will be used for rescue pain treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective transtibial amputation for peripheral vascular disease
* age over 18 years
* American Society of Anaesthesiology status II to IV

Exclusion Criteria:

* contraindication to peripheral regional anesthesia
* psychiatric disease
* pregnancy or breastfeeding status
* amputation for tumour surgery
* traumatic amputation
* inability to give written and informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Point prevalence of chronic phantom limb pain | 12 months after amputation

CONTACTS AND LOCATIONS:
Overall Officials: Markus Hollmann, MD PhD, Study Chair — Dept. of Anaesthesiology, Academic Medical Center / University of Amsterdam, The Netherlands; Philipp Lirk, MD PhD, Principal Investigator — Dept. of Anaesthesiology, Academic Medical Center / University of Amsterdam, The Netherlands
Locations (9):
- Massachusetts General Hospital, Dept. of Anesthesiology, Perioperative and Pain Medicine, Boston, Massachusetts, United States
- Austria (2):
  - General Hospital Klagenfurt, Klagenfurt, Carinthia
  - Innsbruck Medical University Hospital, Innsbruck, Tyrol
- Ziekenhuis Oost Limburg, Genk, Limburg, Belgium
- Netherlands (4):
  - Academic Medical Center, University of Amsterdam, Amsterdam, North Holland
  - Westfriesgasthuis, Hoorn, North Holland
  - Erasmus Medical Center, Rotterdam, North Holland
  - Canisius Wilhelmus Ziekenhuis, Nijmegen
- Valencia University Hospital, Valencia, Spain

REFERENCES:
- [Background] Ypsilantis E, Tang TY. Pre-emptive analgesia for chronic limb pain after amputation for peripheral vascular disease: a systematic review. Ann Vasc Surg. 2010 Nov;24(8):1139-46. doi: 10.1016/j.avsg.2010.03.026. PMID 20800987
- [Background] Rathmell JP, Kehlet H. Do we have the tools to prevent phantom limb pain? Anesthesiology. 2011 May;114(5):1021-4. doi: 10.1097/ALN.0b013e31820fc80d. No abstract available. PMID 21383618